CLINICAL TRIAL: NCT05760027
Title: Effect of Plyometric Exercise on Stability in Professional Indoor Soccer Players: A Pilot Study
Acronym: PESF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Inmaculada Ruiz Lopez, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: UCAM CE012305
Record Dates: First submitted 2023-02-02; First posted 2023-03-08 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Plyometric Exercises
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The evaluator performing the measurements will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric exercise (Experimental): The group of athletes will perform plyometric stability exercises and their usual exercise for 30 days.
  Interventions: Other: Plyometric exercise
- Regular exercise (Other): The group of athletes will their usual exercise for 30 days.
  Interventions: Other: Regular exercise

INTERVENTIONS:
Other: Plyometric exercise — The group of athletes will perform plyometric stability exercises and their usual exercise for 30 days.
  Arms: Plyometric exercise
Other: Regular exercise — The group of athletes will perform their usual exercise for 30 days.
  Arms: Regular exercise

SUMMARY:
A program is proposed for two groups of professional indoor soccer players where the effect of plyometric exercises on body stability will be evaluated on a stabilometric platform.

DETAILED DESCRIPTION:
A program is proposed for two groups of professional indoor soccer players where the effect of plyometric exercises on body stability will be evaluated on a stabilometric platform.

Four evaluations will be carried out. An initial measurement before the beginning of the first intervention phase (Visit 1), after the intervention (Visit 2; day 30), after a 15-day washout period (Visit 3; day 45) and after the second intervention phase (Visit 4; day 75).

ELIGIBILITY:
Inclusion Criteria:

* Professional soccer player in the first division of the National Soccer League (LNFS).
* Age between 18 and 35 years old.
* BMI between 18 and 32 Kg/m2.

Exclusion Criteria:

* Serious or terminal illness.
* Participants with pain associated with chronic conditions.
* Participants with body mass index above 32 kg/m2.
* Inability to understand the informed consent.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Balance Phase 1 | Baseline and end of each intervention [Day 0 and day 30].
  Measurement of the balance measured as a percentage by pressure platform of professional indoor soccer players.
Balance Phase 2 | Baseline and end of each intervention [Day 45 and day 75].
  Measurement of the balance measured as a percentage by pressure platform of professional indoor soccer players.

SECONDARY OUTCOMES:
Flexibility | Baseline and end of each intervention [Day 0 and day 30].
  Flexibility will be measured with goniometer.
Flexibility | Baseline and end of each intervention [Day 45 and day 75].
  Flexibility will be measured with goniometer.
Flexibility | Baseline and end of each intervention [Day 0 and day 30].
  Flexibility will be measured with Lunge test.
Flexibility | Baseline and end of each intervention [Day 45 and day 75].
  Flexibility will be measured with Lunge test.
Number of injuries | Baseline and end of each intervention [Day 0 and day 30].
  The number of lesions will be collected during the course of the study.
Number of injuries | Baseline and end of each intervention [Day 45 and day 75].
  The number of lesions will be collected during the course of the study.
Lower limb pain | Baseline and end of each intervention [Day 0 and day 30].
  Pain intensity will be measured with a Visual Analog Score (minimum value 0 - Maximum value 10). Higher values indicate a greater degree of pain
Lower limb pain | Baseline and end of each intervention [Day 45 and day 75].
  Pain intensity will be measured with a Visual Analog Score (minimum value 0 - Maximum value 10). Higher values indicate a greater degree of pain
Anthropometric measurements | Baseline and end of each intervention [Day 0 and day 30].
  Anthropometric variables measured with a TANITA equipment.
Anthropometric measurements | Baseline and end of each intervention [Day 45 and day 75].
  Anthropometric variables measured with a TANITA equipment.

CONTACTS AND LOCATIONS:
Overall Officials: Universidad Católica San Antonio de Murcia Universidad Católica San Antonio de Murcia, Principal Investigator — Universidad Católica San Antonio de Murcia
Locations (1):
- Universidad Católica San Antonio de Murcia, Murcia, Spain